CLINICAL TRIAL: NCT00060762
Title: Effectiveness of Psychological Treatments for BED
Brief Title: Effectiveness of Binge Eating Disorder Treatments
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH063863 (NIH); R01MH063863 (NIH); DSIR 83-ATAS
Record Dates: First submitted 2003-05-12; First posted 2003-05-13 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Eating Disorders
Keywords: Weight Loss
MeSH Terms: conditions — Feeding and Eating Disorders; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Interpersonal Therapy (Experimental): Interpersonal Therapy is a psychotherapy aimed at resolving interpersonal difficulties
  Interventions: Behavioral: Interpersonal Therapy
- Behavioral Weight Loss Treatment (Active Comparator): Behavioral Weight Loss Treatment is aimed solely at weight loss, however it has been shown to decrease binge eating
  Interventions: Behavioral: Behavioral Weight Loss Treatment
- Guided Self Help (Active Comparator): Guided Self-Help is a brief psychotherapy based on cognitive-behavioral treatment
  Interventions: Behavioral: Guided Self Help

INTERVENTIONS:
Behavioral: Interpersonal Therapy — 20 sessions of interpersonal therapy were provided over a 6-month period
  Other Names: IPT
  Arms: Interpersonal Therapy
Behavioral: Behavioral Weight Loss Treatment — 20 sessions of behavioral weight loss treatment were provided over a 6-month period
  Other Names: BWL; Weight loss treatment
  Arms: Behavioral Weight Loss Treatment
Behavioral: Guided Self Help — 10 sessions of guided self help were provided over a 6-month period
  Other Names: GSH
  Arms: Guided Self Help

SUMMARY:
This study will evaluate the long-term effectiveness of interpersonal psychotherapy, behavioral weight loss interventions, and guided self help treatments in treating binge eating disorder (BED).

DETAILED DESCRIPTION:
BED is a serious condition that is associated with psychiatric comorbidity, psychosocial impairment, and obesity. Interpersonal psychotherapy (IPT), behavioral weight loss (BWL) interventions, and guided self help (GSH) treatments for BED have been evaluated, but the safest and most effective treatment has not yet been identified. This study will determine which of these three treatments is most effective in treating BED.

Participants are stratified by negative affect subtype and are randomly assigned for 6 months to one of three treatment groups: IPT, BWL, or GSH. IPT focuses on current interpersonal problems which are hypothesized to increase negative affect and lead to binge eating. BWL interventions involve the adoption of weight loss inducing behaviors. GSH is a shortened version of cognitive behavioral therapy that focuses directly on eating behavior. IPT and BWL patients have 20 treatment sessions; those receiving GSH have 10 sessions. Assessments are made pre-treatment, post-treatment, and at 6, 12, 18, and 24 months after treatment is complete.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for Binge Eating Disorder
* Body Mass Index (BMI) between 27 and 45

Exclusion criteria:

* Body Mass index > 45
* Current psychosis
* Current bipolar disorder
* Alcohol or drug dependence within last 6-months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2002-04; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Binge eating | Pre-treatment, 6, 12, and 24-months
  Rate of binge eating

SECONDARY OUTCOMES:
Eating disorder psychopathology | pre-treatment, 6, 12, 24 months
  Assessed by the Eating Disorder Examination

CONTACTS AND LOCATIONS:
Overall Officials: William S Agras, MD, Study Director — Stanford University
Locations (3):
- United States (3):
  - W. Stewart Agras, Stanford, California
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers University Eating Disorder Clinic, Piscataway, New Jersey

REFERENCES:
- [Result] Wilson GT, Wilfley DE, Agras WS, Bryson SW. Psychological treatments of binge eating disorder. Arch Gen Psychiatry. 2010 Jan;67(1):94-101. doi: 10.1001/archgenpsychiatry.2009.170. PMID 20048227